CLINICAL TRIAL: NCT03706339
Title: Reducing Blood Loss During Cesarean Section With Intravenous Versus Topical Tranexamic Acid: a Double-blinded Randomized Placebo-controlled Trial
Brief Title: Reducing Blood Loss During Cesarean Section by Topical Versus IV Tranexamic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/278/7/18
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: patients were allocated to one of three groups after induction of general anesthesia and immediately prior to the operation and just before skin incision. they received 1-gram tranexamic acid (10 ml) in 100 ml saline infusion or placebo (110 normal saline) by slow intravenous injection at an approximate rate of 1 mL per min. Throughout the operation irrigation was done by 60 ml of (2g tranexamic acid (10 ml) diluted in 100 ml of sodium chloride 0.9%) or placebo ( 60 ml of sodium chloride 0.9%.).At the end of operation another dose of 60 ml of (1g tranexamic acid (10 ml) diluted in 50 ml of sodium chloride 0.9%) or placebo ( 60 ml of sodium chloride 0.9%.) was left intraabdominal
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal saline arm group (Placebo Comparator): they received 110 ml saline infusion or placebo (110 normal salines) by slow intravenous injection at an approximate rate of 1 mL per min plus Throughout the operation irrigation was done by120 ml saline
  Interventions: Other: normal saline arm group
- intravenous tranexamic acid group (Active Comparator): 1 gm tranexamic acid (2 ampoules of Capron 500 mg /5 ml; Cairo, Egypt) intravenous just before skin incision plus100 ml normal saline IV just before skin incision plus topical application of 120 ml normal saline applied on the pelvic bed after Cesarean hysterectomy
  Interventions: Drug: intravenous tranexamic acid
- Topical tranexamic acid group (Experimental): 2 gm topical tranexamic acid ( 4 ampoules of Capron 500 mg/5 ml applied typically) in 100 ml normal saline applied on the placental bed after Cesarean section plus110 ml normal saline IV just before skin incision
  Interventions: Drug: Topical tranexamic acid

INTERVENTIONS:
Other: normal saline arm group — 110 ml normal saline IV just before skin incision plus topical application of 120 ml normal saline applied on the placental bed during Cesarean section
  Other Names: placebo comparator
  Arms: normal saline arm group
Drug: intravenous tranexamic acid — 1 gm tranexamic acid (2 ampoules of Capron 500 mg /5 ml; Cairo, Egypt) intravenous just before skin incision plus110 ml normal saline IV just before skin incision plus topical application of 120 ml normal saline applied on the pelvic bed during cesarean section
  Other Names: active comparator
  Arms: intravenous tranexamic acid group
Drug: Topical tranexamic acid — 2 gm topical tranexamic acid ( 4 ampoules of Capron 500 mg/5 ml applied typically) in 120 ml normal saline applied on the pelvic bed during cesarean section plus110 ml normal saline IV just before skin incision
  Other Names: active comparator
  Arms: Topical tranexamic acid group

SUMMARY:
Tranexamic (TXA)acid is an inexpensive, antifibrinolytic drug long used to control bleeding due to surgery, menorrhagia, or trauma. Additionally, tranexamic acid has been shown to reduce bleeding during cesarean delivery as well as the need for additional uterotonic agents, albeit to a minimal degree. However, previous studies have been performed only in women with a standard risk for postpartum hemorrhage( PPH) and have not focused on assessing the effects of tranexamic acid in high-risk women. The aim of this study is to evaluate the efficacy of IV versus topical application of tranexamic acid in reducing blood loss during and after elective C.S. The Research Question Is topical application of Tranexamic acid effective in reducing blood loss during and after an elective Caesarean section? The Research Hypothesis the TXA could be able to reduce blood loss during and after elective Caesarean section. The null hypothesis will, therefore, state that: There will be no difference between topical and IV TXA and placebo in reducing blood loss during and after elective Caesarean section.

DETAILED DESCRIPTION:
patients were allocated to one of three groups after induction of general anesthesia and immediately prior to the operation and just before skin incision. they received 1-gram tranexamic acid (10 ml) in 100 ml saline infusion or placebo (110 normal saline) by slow intravenous injection at an approximate rate of 1 mL per min. Throughout the operation, irrigation was done by 60 ml of (2g tranexamic acid (10 ml) diluted in 100 ml of sodium chloride 0.9%) or placebo ( 60 ml of sodium chloride 0.9%.).At the end of operation, another dose of 60 ml of (1g tranexamic acid (10 ml) diluted in 50 ml of sodium chloride 0.9%) or placebo ( 60 ml of sodium chloride 0.9%.) was left intraabdominal

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women with a single term fetus scheduled for elective cesarean section who will be at risk of postpartum hemorrhage

Exclusion Criteria:

* Patients with a cardiac, hepatic, renal or thromboembolic disease. ,
* patients with the high possibility of the morbid adherent placenta,
* known coagulopathy and
* those presented with severe antepartum hemorrhage
* refuse to participate

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with a single term fetus scheduled for an elective Cesarean section
Enrollment: 450 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
intraoperative blood loss | during the operation
  measures the intraoperative blood loss by direct and gravimetric methods

SECONDARY OUTCOMES:
postoperative blood loss | 24 hours postoperative
  measurement the intraoperative blood loss by direct and gravimetric methods
need of blood transfusion | 24 hours postoperative
  number of unites of blood transfusion
need of uterotonic | during operation
  misoprostol,oxytocin etc
change in hemoglobin | Baseline and 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No